CLINICAL TRIAL: NCT06154369
Title: Promoting Mental Health and Wellbeing Among Post-secondary Students With the Joypop App: A Randomized Controlled Trial
Brief Title: JoyPop Mobile Mental Health App With Post-Secondary Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lakehead University (Other)
Responsible Party: Principal Investigator, Aislin Mushquash, Associate Professor, Lakehead University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 100251
Record Dates: First submitted 2023-11-23; First posted 2023-12-04 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Emotion Regulation; Depression; Anxiety; Stress; Well-Being, Psychological
MeSH Terms: conditions — Emotional Regulation; Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: A pragmatic, randomized controlled trial will be used. Participants will be randomly allocated in a 1:1 ratio to the control (no intervention) or intervention (JoyPop) condition. Block randomization (block size of 8) will be used to randomly assign participants to each condition.
Who Masked: Investigator
Masking Description: Given the nature of this trial, it will not be possible to blind participants to their allocation. As measures are self report, blinding of outcome measures is also not possible. Protect against bias will occur by blinding investigators to condition (i.e., only staff directly managing participants will be unblinded).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- JoyPop (Experimental): Participants will receive access to the Joypop app for 8 weeks.
  Interventions: Behavioral: JoyPop
- No Intervention (No Intervention): No intervention will be offered. After 8 weeks in the control condition, participants will be offered access to the JoyPop app.

INTERVENTIONS:
Behavioral: JoyPop — Participants will be asked to use the app at least twice daily for the first 4 weeks with no further instructions on feature usage or time spent using the app.
  Arms: JoyPop

SUMMARY:
Students within post-secondary education settings are experiencing increasing stress, distress, and mental health difficulties. Many post-secondary education settings have identified student mental health and wellbeing as a priority and yet are struggling to adequately meet the needs of students. This has led to exploring whether technology can be used to help promote mental health and wellbeing among students. The JoyPop app is one mobile mental health app with a growing evidence base. It was developed to support improved emotion regulation - a key challenge among students struggling with distress and mental health difficulties. Using a randomized controlled trial (RCT) design, the primary objective of this research is to determine the effectiveness of the JoyPop app in improving emotion regulation among post-secondary students when compared to no intervention. The secondary objectives are to: (1) Assess change in mental health, wellbeing, and resilience between students in each condition to better understand the app's broader impact; (2) Conduct an economic analysis to determine whether receiving the app reduces other health service use and associated costs; (4) Assess students' perspective on the quality of the JoyPop app.

DETAILED DESCRIPTION:
Students within post-secondary education settings are presented with many exciting opportunities and challenges. However, this is a time when many students experience increasing stress, distress, and mental health difficulties. Many post-secondary education settings have identified student mental health and wellbeing as a priority and yet are struggling to adequately meet the needs of students. This has led to exploring whether technology can be used to help promote mental health and wellbeing among students. Mobile mental health applications (apps) are of particular interest given students' access and use of mobile devices. Despite the promise of mobile mental health apps, significant gaps exist between the growing number of apps available in the public domain and empirical demonstration of the beneficial impacts of apps for users.

The JoyPop app is one mobile mental health app with a growing evidence base. It was developed to support improved emotion regulation - a key challenge among students struggling with distress and mental health difficulties. Of the apps that address emotion regulation, most have not been evaluated, are narrow in scope, or have only been evaluated among non-diverse adult populations. The JoyPop app includes a broader focus, and this research is unique given its focus on rigorously evaluating the JoyPop app as a tool for students within post-secondary settings.

Using a randomized controlled trial (RCT) design, the primary objective is to determine the effectiveness of the JoyPop app in improving emotion regulation among post-secondary students when compared to no intervention. The secondary objectives are to: (1) Assess change in mental health, wellbeing, and resilience between students in each condition to better understand the app's broader impact; (2) Conduct an economic analysis to determine whether receiving the app reduces other health service use and associated costs; (4) Assess students' perspective on the quality of the JoyPop app.

ELIGIBILITY:
Inclusion Criteria:

* Post-secondary student
* Between 18-25 years old
* Speak/read fluently in English
* Available to attend a virtual or in-person orientation session
* In order to download the JoyPop app, participants will need access to an iOS device (e.g., iPhone, iPad). Refurbished iPhones containing just the JoyPop app may be provided to participants to use for the duration of the trial if they do not have access to their own

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2023-11-22 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Change in emotion regulation (overall) | Difficulties in Emotion Regulation Scale - Short Form will be administered at baseline (pre), after 2 weeks (mid), after 4 weeks (post) and after 8 weeks (follow up)
  Emotion regulation will be assessed with the Difficulties in Emotion Regulation Scale - Short Form. Total scores range from 18 to 90 with higher scores indicating greater difficulties in emotion regulation.
Change in emotion regulation (strategies) | Difficulties in Emotion Regulation Scale - Short Form will be administered at baseline (pre), after 2 weeks (mid), after 4 weeks (post) and after 8 weeks (follow up)
  Emotion regulation strategies will be assessed with the Difficulties in Emotion Regulation Scale - Short Form strategies subscale. Total scores range from 3 to 15 with higher scores indicating greater difficulties.
Change in emotion regulation (non-acceptance) | Difficulties in Emotion Regulation Scale - Short Form will be administered at baseline (pre), after 2 weeks (mid), after 4 weeks (post) and after 8 weeks (follow up)
  Emotion regulation strategies will be assessed with the Difficulties in Emotion Regulation Scale - Short Form non-acceptance subscale. Total scores range from 3 to 15, with higher scores indicating greater difficulties.
Change in emotion regulation (impulse) | Difficulties in Emotion Regulation Scale - Short Form will be administered at baseline (pre), after 2 weeks (mid), after 4 weeks (post) and after 8 weeks (follow up)
  Emotion regulation strategies will be assessed with the Difficulties in Emotion Regulation Scale - Short Form impulse subscale. Total scores range from 3 to 15, with higher scores indicating greater difficulties.
Change in emotion regulation (goals) | Difficulties in Emotion Regulation Scale - Short Form will be administered at baseline (pre), after 2 weeks (mid), after 4 weeks (post) and after 8 weeks (follow up)
  Emotion regulation strategies will be assessed with the Difficulties in Emotion Regulation Scale - Short Form impulse subscale. Total scores range from 3 to 15, with higher scores indicating greater difficulties.
Change in emotion regulation (awareness) | Difficulties in Emotion Regulation Scale - Short Form will be administered at baseline (pre), after 2 weeks (mid), after 4 weeks (post) and after 8 weeks (follow up)
  Emotion regulation strategies will be assessed with the Difficulties in Emotion Regulation Scale - Short Form awareness subscale. Total scores range from 3 to 15, with higher scores indicating greater difficulties.
Change in emotion regulation (clarity) | Difficulties in Emotion Regulation Scale - Short Form will be administered at baseline (pre), after 2 weeks (mid), after 4 weeks (post) and after 8 weeks (follow up)
  Emotion regulation strategies will be assessed with the Difficulties in Emotion Regulation Scale - Short Form clarity subscale. Total scores range from 3 to 15, with higher scores indicating greater difficulties.

SECONDARY OUTCOMES:
Change in psychological distress | Depression Anxiety and Stress Scale 21 will be administered at baseline (pre), after 2 weeks (mid), after 4 weeks (post) and after 8 weeks (follow up)
  Psychological distress will be assessed with the total score for all items on the Depression Anxiety and Stress Scale 21. Total scores range from 0 to 63, with higher scores indicating greater psychological distress.
Change in depressive symptoms | Depression Anxiety and Stress Scale 21 will be administered at baseline (pre), after 2 weeks (mid), after 4 weeks (post) and after 8 weeks (follow up)
  Depressive symptoms will be assessed with the Depression subscale of the Depression Anxiety and Stress Scale 21. Total scores range from 0 to 21, with higher scores indicating greater depressive symptoms.
Change in anxious symptoms | Depression Anxiety and Stress Scale 21 will be administered at baseline (pre), after 2 weeks (mid), after 4 weeks (post) and after 8 weeks (follow up)
  Anxious symptoms will be assessed with the Anxiety subscale of the Depression Anxiety and Stress Scale 21. Total scores range from 0 to 21 with higher scores indicating greater anxious symptoms.
Change in stress | Depression Anxiety and Stress Scale 21 will be administered at baseline (pre), after 2 weeks (mid), after 4 weeks (post) and after 8 weeks (follow up)
  Stress will be assessed with the Stress subscale of the Depression Anxiety and Stress Scale 21. Total scores range from 0 to 21, with higher scores indicating greater stress.
Change in mental health symptoms | General Health Questionnaire 12 will be administered at baseline (pre), after 2 weeks (mid), after 4 weeks (post), and after 8 weeks (follow up)
  Mental health symptoms will be assessed with the total score for all items on the General Health Questionnaire 12. Total scores range from 0 to 36 with higher scores indicating greater distress.
Change in mental well-being | Warwick Edinburgh Mental Wellbeing Scale will be administered at baseline (pre), after 2 weeks (mid), after 4 weeks (post), and after 8 weeks (follow up)
  Mental well-being will be assessed with the total score for all items on the 14-item Warwick Edinburgh Mental Wellbeing Scale. Total scores range from 14 to 70 with a higher score indicating greater mental well-being.
Change in resilience | Connor-Davidson Resilience Scale-10 will be administered at baseline (pre), after 2 weeks (mid), after 4 weeks (post), and after 8 weeks (follow up)
  Resiliency will be assessed with the total score for all items on the Conner-Davidson Resilience Scale-10. Total scores range from 0 to 40 with higher scores indicating greater resiliency.

OTHER OUTCOMES:
Self-reported healthcare utilization | Service utilization measure will be administered at baseline (pre), after two weeks (mid), after four weeks (post), and after 8 weeks (follow up)
  Service utilization will be assessed with 5 items asking about frequency of healthcare services accessed over the prior 2 weeks. Response options are open-ended and will be analyzed individually and as a total score across service types.
App quality (overall) | User Version of the Mobile Application Rating Scale will be administered to the intervention group after 4 weeks (post)
  App quality (overall) will be assessed with the User Version of the Mobile Application Rating Scale. Total scores range from 1 to 5, with higher scores indicating greater quality.
App quality (engagement) | User Version of the Mobile Application Rating Scale will be administered to the intervention group after 4 weeks (post)
  App quality (engagement) will be assessed with the Engagement subscale of the User Version of the Mobile Application Rating Scale. Total scores range from 1 to 5, with higher scores indicating greater quality (engagement).
App quality (functionality) | User Version of the Mobile Application Rating Scale will be administered to the intervention group after 4 weeks (post)
  App quality (functionality) will be assessed with the Functionality subscale of the User Version of the Mobile Application Rating Scale. Total scores range from 1 to 5, with higher scores indicating greater quality (functionality).
App quality (aesthetics) | User Version of the Mobile Application Rating Scale will be administered to the intervention group after 4 weeks (post)
  App quality (aesthetics) will be assessed with the Aesthetics subscale of the User Version of the Mobile Application Rating Scale. Total scores range from 1 to 5, with higher scores indicating greater quality (aesthetics).
App quality (information) | User Version of the Mobile Application Rating Scale will be administered to the intervention group after 4 weeks (post)
  App quality (information) will be assessed with the Information subscale of the User Version of the Mobile Application Rating Scale. Total scores range from 1 to 5, with higher scores indicating greater quality (information).
App quality (subjective) | User Version of the Mobile Application Rating Scale will be administered to the intervention group after 4 weeks (post)
  App quality (subjective) will be assessed with the App Subjective Quality items of the User Version of the Mobile Application Rating Scale. Items will be assessed individually and as a total score (range from 1 to 5), with higher scores indicating greater quality (subjective).
App quality (perceived impact) | User Version of the Mobile Application Rating Scale will be administered to the intervention group after 4 weeks (post)
  App quality (perceived impact) will be assessed with the Perceived Impact subscale of the User Version of the Mobile Application Rating Scale. Items will be assessed individually and as a total score (range from 1 to 5), with higher scores indicating greater quality (perceived impact).

CONTACTS AND LOCATIONS:
Locations (1):
- Lakehead University, Thunder Bay, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] MacIsaac A, Mann V, Toombs E, Schmidt F, Olthuis JV, Stewart SH, Newton A, Ohinmaa A, Mushquash AR. Promoting mental health and wellbeing among post-secondary students with the JoyPop app: study protocol for a randomized controlled trial. Trials. 2024 Sep 2;25(1):576. doi: 10.1186/s13063-024-08424-y. PMID 39223596